CLINICAL TRIAL: NCT04923100
Title: Therapeutic Effect of New Biologics in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021ZSLYEC-066
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Treatment Side Effects
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — intestinal mucosa biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New types of biologics have brought advantages in therapy strategies for Crohn's disease. However, clinical data evaluating their efficacy and adverse in China is lacking. We aimed to evaluate the short-term and long-term therapeutic effect as well as drug adverse of Ustekinumab (UST) and Vedolizumab (VED). Besides, we aim to figure out the independent factors predicting the effectiveness of new biologics. Relations between drug exposure (trough concentration and antibody concentration) and therapeutic efficacy are study in-depth by this retrospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients with confirmed diagnosis of Crohn's disease and administration of new type biologics.

Exclusion Criteria:

* loss of follow-up, incomplete clinical data, without confirmed diagnosis

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult patients with confirmed diagnosis of Crohn's disease and administration of new type biologics
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
endoscopic remission | short-time efficacy (16-20 weeks or 24 weeks) and long-term efficacy (52~54weeks)
  Endoscopic remission referred to those with simple endoscopic score for Crohn's disease (SES-CD)≤2

SECONDARY OUTCOMES:
clinical remission | short-time efficacy (16-20 weeks or 24 weeks) and long-term efficacy (52~54weeks)
  Clinical remission was defined as Crohn's disease activity index (CDAI) below 150
clinical response | short-time efficacy (16-20 weeks or 24 weeks) and long-term efficacy (52~54weeks)
  endoscopic response referred to those with a reduction of SES-CD > 50% baseline
endoscopic response | short-time efficacy (16-20 weeks or 24 weeks) and long-term efficacy (52~54weeks)
  endoscopic response referred to those with a reduction of SES-CD > 50% baseline

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yao J, Peng X, Zhong Y, Su T, Bihi A, Zhao J, Liu T, Wang W, Hu P, Zhang M, Zhi M. Extra intravenous Ustekinumab reinduction is an effective optimization strategy for patients with refractory Crohn's disease. Front Med (Lausanne). 2023 Jul 24;10:1105981. doi: 10.3389/fmed.2023.1105981. eCollection 2023. PMID 37554510
- [Derived] Yao JY, Zhang M, Wang W, Peng X, Zhao JZ, Liu T, Li ZW, Sun HT, Hu P, Zhi M. Ustekinumab trough concentration affects clinical and endoscopic outcomes in patients with refractory Crohn's disease: a Chinese real-world study. BMC Gastroenterol. 2021 Oct 18;21(1):380. doi: 10.1186/s12876-021-01946-8. PMID 34663208